CLINICAL TRIAL: NCT01352793
Title: A Phase 3, Randomized, Active-controlled, Observer-blinded Trial To Assess The Safety And Tolerability Of A Meningococcal Serogroup B Bivalent Recombinant Lipoprotein (rlp2086) Vaccine Given In Healthy Subjects Aged Greater Than Or Equal To 10 To Less Than 26 Years
Brief Title: A Global Phase 3 Safety Study of 120 mcg rLP2086 Vaccine in Adolescents and Young Adults Aged 10 to 25 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1971014; 2009-015198-11 (EudraCT Number); 6108A1-3003 (Other: Alias Study Number)
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Meningitis, Meningococcal
Keywords: phase 3 safety study; 5700 healthy subjects; 3 vaccine doses at month 0; 2; and 6; control HAV/saline/HAV
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rLP2086 vaccine (Experimental): rLP2086 vaccine
  Interventions: Biological: rLP2086 vaccine
- control (Other): The control treatment will be HAVRIX vaccine at month 0 and 6 and a normal saline injection at month 2.
  Interventions: Biological: control

INTERVENTIONS:
Biological: rLP2086 vaccine — 120 mcg, 3 doses, at month 0, 2, and 6.
  Arms: rLP2086 vaccine
Biological: control — HAVRIX: 720 EL.U. or 1440 EL.Ul, 2 doses, at month 0 and 6. Placebo: normal saline injection, 1 dose, at month 2.
  Arms: control

SUMMARY:
A multicenter phase 3 safety trial in which 5,700 subjects will be assigned in a 2:1 ratio to receive 120 μg rLP2086 vaccine in a 0, 2, 6 month schedule or control. The control group will receive HAVRIX vaccine at month 0 and 6 and saline at month 2.

All subjects will be followed for 6 months after the last vaccination to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 10 to 25 years.

Exclusion Criteria:

* Previous vaccination with Hepatitis A virus vaccine
* Previous vaccination with investigational meningococcal B vaccine
* History of culture-proven N. meningitidis serogroup B disease
* Any neuroinflammatory or autoimmune condition
* Any immune defect that would prevent an effective response to the study vaccine

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5715 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (85):
- United States (39):
  - Accelovance,Inc., Huntsville, Alabama
  - Clinical Research Advantage, Inc. / East Valley Family Physicians, PLC, Chandler, Arizona
  - Clinical Research Advantage, Inc/ East Valley Family Physicians, PLC, Chandler, Arizona
  - Cassidy Medical Group/Clinical Research Advantage, Tempe, Arizona
  - Clinical Research Advantage, Inc. / East Valley Family Physicians, PLC, Tempe, Arizona
  - Clinical Research Advantage, Inc./Prairie Fields Family Medicine, PC Administrative/Mailing Address, Tempe, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Accelovance. Inc, San Diego, California
  - Benchmark Research, San Francisco, California
  - Cassidy Medical Group/Clinical Research Advantage, Vista, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - Accelovance, Melbourne, Florida
  - Miami Research Associates, South Miami, Florida
  - Accelovance,Inc., Mishawaka, Indiana
  - Clinical Research Advantage,Inc/Ridge Family Practice, Council Bluffs, Iowa
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Clinical Research Advantage, Inc./ Pediatric Partners, LLC Additional Site-No IP, Fremont, Nebraska
  - Prairie Fields Family Medicine/Clinical Research Advantage, Fremont, Nebraska
  - Rochester Clinical Research, Inc., Rochester, New York
  - Rapid Medical Research. Inc., Cleveland, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Bristol, Bristol, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Research Across America, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Research Across America, Katy, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - J. Lewis Research, Inc. - Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Pediatric Research of Charlottesville, Charlottesville, Virginia
- Australia (5):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - AusTrials Pty Ltd, Sherwood, Queensland
  - Vaccinology and Immunology Research Trials Unit (VIRTU), Discipline of Paediatrics, North Adelaide, South Australia
  - Telethon Institute for Child Health Research, Subiaco
- Chile (5):
  - Centro De Investigacion Clinica Del Sur, Temuco, Región de la Araucanía
  - Cesfam Dr. Jose Symon Ojeda, Conchalí, Santiago Metropolitan
  - Hospital Clinico de la Pontificia Universidad Catolica de Chile/, Santiago, Santiago Metropolitan
  - Centro de Estudios de Vacunas, CESFAM Gabriela Mistral, Santiago, Santiago Metropolitan
  - Hospital Luis Calvo Mackenna, Santiago
- Czechia (5):
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Ordinace praktickeho lekare pro deti a dorost, Pilsen
  - Ordinace praktickeho lekare pro deti a dorost, Prague
  - Prakticky Lekar Pro Deti a Mladez, Týnec nad Sázavou
- Aarhus Universitetshospital, Skejby, Aarhus N, Denmark
- Estonia (4):
  - Eraarst Kersti Veidrik Ou, Rakvere
  - Innomedica OU, Tallinn
  - Merekivi Perearstid OU, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
- Finland (3):
  - Pori Vaccine Research Clinic, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Germany (4):
  - Clinical Trial Center North, Hamburg
  - Clinical Trial Center North GmbH & Co.KG, Hamburg
  - Bernhard Nocht Centre for Clinical Trials (BNCCT), Hamburg
  - Juliusspital Wuerzburg, Würzburg
- Lithuania (5):
  - JSC "InMedica", Kaunas
  - Saules Family Medicine Centre, Kaunas
  - Kaunas Clinical Hospital, Public Institution, Clinic of Infectious Diseases, Kaunas
  - LITHUANIAN HEALTH SCIENCE UNIVERSITY HOSPITAL, CLINIC of FAMILY MEDICINE, Kaunas
  - Centro poliklinika, Public Institution, Vilnius
- Poland (10):
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow, Poland
  - Prywatny Gabinet Lekarski Dr.n.med.Jerzy Brzostek, Dębica
  - Hanna Czajka Indywidualna Specjalistyczna Praktyka Lekarska, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Oddzial Pediatryczny, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego Alina Grocka-Wlazlak, Oborniki Śląskie
  - Specjalistyczny Zespol Opieki Zdrowotnej nad Matka i Dzieckiem w Poznaniu, Poznan
  - NZLA Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - NZOZ Nasz Lekarz, Torun
  - Szpital im. Sw. Jadwigi Slaskiej, Oddzial Pediatryczny, Trzebnica
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Spain (2):
  - Instituto Hispalense de Pediatria, Seville, Sevilla
  - Clinicas Universitarias. Universidad Catolica de Valencia San Vicente Martir, Valencia, Valencia
- Sweden (2):
  - Vaccinenheten Barn- och ungdomsmedicinska kliniken, Malmo, SE
  - Norrlands Universitetssjukhus, Institution för Pediatrik, Umeå

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971014&StudyName=A%20Global%20Phase%203%20Safety%20Study%20of%20120%20mcg%20rLP2086%20Vaccine%20in%20Adolescents%20and%20Young%20Adults%20Aged%2010%20to%2025%20Years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5712 participants in 12 countries were enrolled in this study. Of these, 8 participants were randomized but did not receive study vaccination.
Groups:
- Group 1: rLP2086: Randomized to receive Neisseria meningitidis serogroup B (MnB) bivalent recombinant lipoprotein 2086 (rLP2086) vaccine on a 0, 2-, 6-month schedule
- Group 2: HAV/Saline/HAV: Randomized to receive hepatitis A virus (HAV) vaccine (Havrix) on a 0-, 6- month schedule and normal saline on 2-month
Period: Overall Study
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Started | 3804 | 1908
Vaccination 1 | 3796 | 1908
Vaccination 2 | 3530 | 1806
Vaccination 3 | 3314 | 1710
Completed | 3219 | 1663
Not Completed | 585 | 245
Not completed — Lost to Follow-up | 289 | 125
Not completed — Withdrawal by Subject | 120 | 55
Not completed — Protocol Violation | 44 | 23
Not completed — Adverse Event | 44 | 10
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 26 | 8
Not completed — Other | 25 | 7
Not completed — Medication error | 2 | 2
Not completed — Death | 1 | 0
Not completed — Randomized but not vaccinated | 8 | 0
Not completed — No longer meets eligibility criteria | 25 | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV | Total
Number analyzed (Participants) | 3804 | 1908 | 5712
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.4 (4.6) | 17.4 (4.6) | 17.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1962 | 994 | 2956
  Male | 1842 | 914 | 2756

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) Throughout the Study
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly.
Time Frame: Vaccination 1 up to 6 months after Vaccination 3
Population: Safety population included all participants who received at least 1 dose of study vaccine (bivalent rLP2086 or HAV vaccine or saline) and had safety information available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants | 1.55 [1.2 to 2.0] | 2.52 [1.9 to 3.3]

2. Primary Outcome: Percentage of Participants With at Least One Medically Attended Adverse Event Within 30 Days After Vaccination 1
Description: A medically attended AE was defined as a non-serious AE that required medical attention.
Time Frame: Within 30 days after Vaccination 1
Population: Vaccination 1 safety population included all participants who received the first dose of study vaccine (bivalent rLP2086 or HAV vaccine) and had safety information available from Vaccination 1 until prior to Vaccination 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants | 7.03 [6.2 to 7.9] | 6.13 [5.1 to 7.3]

3. Primary Outcome: Percentage of Participants With at Least One Medically Attended Adverse Event Within 30 Days After Vaccination 2
Description: A medically attended AE was defined as a non-serious AE that required medical attention.
Time Frame: Within 30 days after Vaccination 2
Population: Vaccination 2 safety population included all participants who received the second dose of study vaccine (bivalent rLP2086 or saline) and had safety information available from Vaccination 2 until prior to Vaccination 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3529 | 1806
percentage of participants | 5.50 [4.8 to 6.3] | 6.09 [5.0 to 7.3]

4. Primary Outcome: Percentage of Participants With at Least One Medically Attended Adverse Event Within 30 Days After Vaccination 3
Description: A medically attended AE was defined as a non-serious AE that required medical attention.
Time Frame: Within 30 days after Vaccination 3
Population: Vaccination 3 safety population included all participants who received the third dose of study vaccine (bivalent rLP2086 or HAV vaccine or saline) and had safety information available from Vaccination 3 to post Vaccination 3 follow-up visit (1 month after Vaccination 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3313 | 1710
percentage of participants | 5.34 [4.6 to 6.2] | 5.50 [4.50 to 6.7]

5. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) During Pre-specified Time Periods
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Here, 'N' signifies those participants who were evaluable for this measure during specified time period.
Time Frame: Within 30 days after Vaccination 1, 2, 3, any vaccination; vaccination phase (Vaccination 1 up to 1 month after Vaccination 3); follow-up phase (1 month up to 6 months after Vaccination 3)
Population: Safety population included all participants who received at least 1 dose of the study vaccine (bivalent rLP2086 or HAV vaccine or saline) and had safety information available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants
  30 days after Vaccination 1 (N=3796, 1908) | 0.18 [0.1 to 0.4] | 0.42 [0.2 to 0.8]
  30 days after Vaccination 2 (N=3529, 1806) | 0.17 [0.1 to 0.4] | 0.44 [0.2 to 0.9]
  30 days after Vaccination 3 (N=3313, 1710) | 0.33 [0.2 to 0.6] | 0.12 [0.0 to 0.4]
  30 days after any vaccination (N=3796, 1908) | 0.61 [0.4 to 0.9] | 0.94 [0.6 to 1.5]
  Vaccination phase (N=3796, 1908) | 1.16 [0.8 to 1.6] | 1.83 [1.3 to 2.5]
  Follow-up phase (N=3400, 1733) | 0.44 [0.2 to 0.7] | 0.87 [0.5 to 1.4]

6. Secondary Outcome: Percentage of Participants With at Least One Medically Attended Adverse Event During Pre-specified Time Periods
Description: A medically attended AE was defined as a non-serious AE that required medical attention.
Time Frame: Within 30 days after any vaccination; vaccination phase (Vaccination 1 up to 1 month after Vaccination 3); follow-up phase (1 month up to 6 months after Vaccination 3); throughout study (Vaccination 1 up to 6 months after Vaccination 3)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants
  30 days after any vaccination (N=3796, 1908) | 14.38 [13.3 to 15.5] | 14.57 [13.0 to 16.2]
  Vaccination phase (N=3796, 1908) | 24.60 [23.2 to 26.0] | 24.53 [22.6 to 26.5]
  Follow-up phase (N=3400, 1733) | 11.24 [10.2 to 12.3] | 11.43 [10.0 to 13.0]
  Throughout study (N=3796, 1908) | 29.00 [27.6 to 30.5] | 29.04 [27.0 to 31.1]

7. Secondary Outcome: Percentage of Participants With at Least One Newly Diagnosed Chronic Medical Condition During Pre-specified Time Periods
Description: A newly diagnosed chronic medical condition was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects. Newly diagnosed chronic medical condition did not include illnesses considered to be temporary conditions. Here, 'N' signifies those participants who were evaluable for this measure during specified time period.
Time Frame: Within 30 days after Vaccination 1, 2, 3, any vaccination; vaccination phase(Vaccination 1 up to 1 month after Vaccination 3); follow-up phase(1 month up to 6 months after Vaccination 3); throughout study(Vaccination 1 up to 6 months after Vaccination 3)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants
  30 days after Vaccination 1 (N=3796, 1908) | 0.21 [0.1 to 0.4] | 0.10 [0.0 to 0.4]
  30 days after Vaccination 2 (N=3529, 1806) | 0.17 [0.1 to 0.4] | 0.33 [0.1 to 0.7]
  30 days after Vaccination 3 (N=3313, 1710) | 0.09 [0.0 to 0.3] | 0.12 [0.0 to 0.4]
  30 days after any vaccination (N=3796, 1908) | 0.45 [0.3 to 0.7] | 0.52 [0.3 to 1.0]
  Vaccination phase (N=3796, 1908) | 1.03 [0.7 to 1.4] | 1.05 [0.6 to 1.6]
  Follow-up phase (N=3400, 1733) | 0.44 [0.2 to 0.7] | 0.52 [0.2 to 1.0]
  Throughout study (N=3796, 1908) | 1.40 [1.0 to 1.8] | 1.52 [1.0 to 2.2]

8. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During Pre-specified Time Periods
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. Here, 'N' signifies those participants who were evaluable for this measure during specified time period.
Time Frame: Within 30 days after Vaccination 1, 2, 3, any vaccination; vaccination phase (Vaccination 1 up to 1 month after Vaccination 3)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants
  30 days after Vaccination 1 (N=3796, 1908) | 31.48 [30.0 to 33.0] | 19.03 [17.3 to 20.9]
  30 days after Vaccination 2 (N=3529, 1806) | 20.37 [19.1 to 21.7] | 12.35 [10.9 to 14.0]
  30 days after Vaccination 3 (N=3313, 1710) | 15.00 [13.8 to 16.3] | 10.76 [9.3 to 12.3]
  30 days after any vaccination (N=3796, 1908) | 43.02 [41.4 to 44.6] | 31.45 [29.4 to 33.6]
  Vaccination phase (N=3796, 1908) | 51.08 [49.5 to 52.7] | 42.51 [40.3 to 44.8]

9. Secondary Outcome: Percentage of Participants With at Least One Immediate Adverse Event (AE) After Each Study Vaccination
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. Any AE that occurred within the first 30 minutes after the administration of study vaccine (bivalent rLP2086, HAV vaccine or saline) was classified as an immediate AE. Here, 'N' signifies those participants who were evaluable for this measure during specified time period.
Time Frame: Within 30 minutes after Vaccination 1, 2, 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
percentage of participants
  Vaccination 1 (N=3796, 1908) | 1.05 [0.8 to 1.4] | 0.84 [0.5 to 1.4]
  Vaccination 2 (N=3529, 1806) | 0.54 [0.3 to 0.8] | 0.06 [0.0 to 0.3]
  Vaccination 3 (N=3313, 1710) | 0.45 [0.3 to 0.7] | 0.41 [0.2 to 0.8]

10. Secondary Outcome: Number of Days Participant Missed School or Work Due to Adverse Events (AEs)
Time Frame: Vaccination 1 up to 1 month after Vaccination 3
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Number analyzed (Participants) | 3796 | 1908
days | 3.0 (7.01) [1 to 110] | 3.0 (9.67) [1 to 136]

ADVERSE EVENTS:
Time Frame: AEs were recorded from Vaccination 1 to 1 month after last vaccination. SAEs, newly diagnosed chronic medical conditions and medically attended adverse events were recorded from Vaccination 1 to 6 months after the last vaccination
Description: SAEs and AEs were grouped by system organ class and summarized. AEs collected on the case report form at each visit (non-systematic assessment).
Arm/Group | Group 1: rLP2086 | Group 2: HAV/Saline/HAV
Serious Adverse Events (participants affected / at risk) | 59/3796 | 48/1908
Other Adverse Events (participants affected / at risk) | 1671/3796 | 640/1908
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 (N=3796) | Group 2: HAV/Saline/HAV (N=1908)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 4
Gastroenteritis (Infections and infestations) | 0 | 3
Peritonsillar abscess (Infections and infestations) | 2 | 1
Meningitis viral (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Meningitis enterococcal (Infections and infestations) | 0 | 1
Meningitis enteroviral (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Salpingitis (Infections and infestations) | 1 | 0
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Central Nervous System germinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1
Demyelination (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Meningism (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 3
Major depression (Psychiatric disorders) | 1 | 1
Substance abuse (Psychiatric disorders) | 2 | 0
Attention deficit or hyperactivity disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 (N=3796) | Group 2: HAV/Saline/HAV (N=1908)
Nausea (Gastrointestinal disorders) | 89 | 33
Vomiting (Gastrointestinal disorders) | 60 | 27
Abdominal pain (Gastrointestinal disorders) | 47 | 32
Diarrhoea (Gastrointestinal disorders) | 42 | 17
Injection site pain (General disorders) | 722 | 149
Pyrexia (General disorders) | 237 | 44
Injection site erythema (General disorders) | 142 | 6
Vaccination site pain (General disorders) | 126 | 9
Fatigue (General disorders) | 82 | 19
Injection site swelling (General disorders) | 84 | 6
Upper respiratory tract infection (Infections and infestations) | 157 | 87
Nasopharyngitis (Infections and infestations) | 149 | 84
Pharyngitis (Infections and infestations) | 75 | 47
Gastroenteritis (Infections and infestations) | 64 | 38
Bronchitis (Infections and infestations) | 65 | 36
Sinusitis (Infections and infestations) | 54 | 33
Urinary tract infection (Infections and infestations) | 50 | 24
Pharyngitis streptococcal (Infections and infestations) | 45 | 22
Tonsillitis (Infections and infestations) | 38 | 21
Viral pharyngitis (Infections and infestations) | 41 | 13
Ligament sprain (Injury, poisoning and procedural complications) | 60 | 30
Contusion (Injury, poisoning and procedural complications) | 50 | 23
Fall (Injury, poisoning and procedural complications) | 38 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 76 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 27
Headache (Nervous system disorders) | 249 | 102
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 83 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.